CLINICAL TRIAL: NCT02559180
Title: Investigator Initiated Observational Study of Intravitreal Aflibercept Injection in Subjects With Diabetic Macular Edema Previously Treated With Ranibizumab or Bevacizumab
Brief Title: Treatment of Diabetic Macular Edema With Aflibercept in Subjects Previously Treated With Ranibizumab or Bevacizumab
Acronym: SwapTwo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rishi Singh (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Rishi Singh, staff surgeon/Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SwapTwo Study
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: Diabetes; Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Diabetes Mellitus | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): aflibercept 2mg given intravitreally every month until resolution of fluid in retina and then continued every 2 months for a total of 24 months of treatment
  Interventions: Drug: aflibercept

INTERVENTIONS:
Drug: aflibercept — aflibercept 2mg given intravitreally every month until resolution of fluid in retina and then continued every 2 months for a total of 24 months of treatment
  Other Names: Eylea

SUMMARY:
Treatment of diabetic macular edema with intravitreal aflibercept in subjects previously treated with intravitreal anti-Vascular endothelial growth factor (VEGF) agents (ranibizumab or bevacizumab)

DETAILED DESCRIPTION:
This study is an investigator initiated interventional study for subjects with diabetic macular edema (DME) that have been previously treated with bevacizumab or ranibizumab. Intravitreal aflibercept 2mg will be given until OCT (ocular coherence tomography) demonstrates an absence of fluid. Continued intravitreal aflibercept 2mg will then take place every 2 months for a total of 24 months of treatment.

This study is an interventional, single arm, investigator initiated study. Subjects will be given 2 mg (0.05 mL or 50 microliters) of intravitreal aflibercept injection (IAI) administered monthly until OCT demonstrates no evidence of fluid as defined by the protocol, followed by 2 mg (0.05 mL) once every 2 months. Each subject will be evaluated for 24 months. Thus, the study duration will be 24 months plus the recruitment period.

Subjects will be evaluated for safety, efficacy as measured by Spectral Domain Optical Coherence Tomography (SDOCT) and best corrected visual acuity (BCVA) using the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) protocol. In additional, fundus photography, fluorescein angiography, and OCT angiography will be performed at baseline, month 6, month 12 and at the final visit.

Only one eye per subject may be enrolled in the study. If a subject's fellow (non-study) eye requires treatment for at study entry, or during the subject's participation in the study, the fellow eye can receive IAI for DME.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Foveal-involving retinal edema secondary to DME based on investigator review of clinical exam and SDOCT with central subfield thickness value of 325 microns by Zeiss Cirrus SD-OCT.
3. E-ETDRS best-corrected visual acuity of: 20/25 to 20/400 in the study eye.
4. History of previous treatment with anti-VEGF with at least 4 injections over the last 6 months.
5. Willing, committed, and able to return for all clinic visits and complete all study related procedures.
6. Able to read, (or, if unable to read due to visual impairment, be read to verbatim by the person administering the informed consent or a family member.) understand and willing to sign the informed consent form.

   -

Exclusion Criteria:

1. Any prior or concomitant therapy with another investigational agent to treat DME in the study eye.
2. Prior panretinal photocoagulation in the study eye within the past 3 months.
3. Prior intravitreal anti-VEGF therapy in the study eye within 30 days of enrollment.
4. Prior systemic anti-VEGF therapy, investigational or FDA-approved, is only allowed up to 3 months prior to first dose, and will not be allowed during the study.
5. Previous treatment with intravitreal aflibercept injection
6. Significant vitreous hemorrhage obscuring view to the macula or the retinal periphery as determined by the investigator on clinical exam
7. Presence of other causes of macular edema, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, choroidal neovascularization, age-related macular degeneration or multifocal choroiditis in the study eye.
8. Presence of macula-threatening traction retinal detachment.
9. Prior vitrectomy in the study eye.
10. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
11. Any history of macular hole of stage 2 and above in the study eye.
12. Any intraocular or periocular surgery within 3 months of Day 1 on the study eye, except lid surgery, which may not have taken place within 1 month of day 1, as long as it's unlikely to interfere with the injection.
13. Uncontrolled glaucoma at baseline evaluation
14. Active intraocular inflammation in either eye.
15. Active ocular or periocular infection in either eye.
16. Any ocular or periocular infection within the last 2 weeks prior to Screening in either eye.
17. Any history of uveitis in either eye.
18. History of corneal transplant or corneal dystrophy in the study eye.
19. Significant media opacities, including cataract, in the study eye which might interfere with visual acuity, assessment of safety, or fundus photography.
20. Any concurrent intraocular condition in the study eye (e.g. cataract) that, in the opinion of the investigator, could require either medical or surgical intervention during the 52 week study period.
21. Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
22. Participation as a subject in any clinical study within the 12 weeks prior to Day 1.
23. Any systemic therapy with an investigational agent in the past 3 months prior to Day 1.
24. Any history of allergy to povidone iodine.
25. Pregnant or breast-feeding women
26. Women of childbearing potential who are unwilling to practice adequate contraception during the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rishi P Singh, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrara N, Davis-Smyth T. The biology of vascular endothelial growth factor. Endocr Rev. 1997 Feb;18(1):4-25. doi: 10.1210/edrv.18.1.0287. No abstract available. PMID 9034784
- [Background] Ferrara N, Houck KA, Jakeman LB, Winer J, Leung DW. The vascular endothelial growth factor family of polypeptides. J Cell Biochem. 1991 Nov;47(3):211-8. doi: 10.1002/jcb.240470305. PMID 1791185
- [Background] Ferrara N. Vascular endothelial growth factor and the regulation of angiogenesis. Recent Prog Horm Res. 2000;55:15-35; discussion 35-6. PMID 11036931
- [Background] Rakic JM, Lambert V, Devy L, Luttun A, Carmeliet P, Claes C, Nguyen L, Foidart JM, Noel A, Munaut C. Placental growth factor, a member of the VEGF family, contributes to the development of choroidal neovascularization. Invest Ophthalmol Vis Sci. 2003 Jul;44(7):3186-93. doi: 10.1167/iovs.02-1092. PMID 12824270
- [Background] Thickett DR, Armstrong L, Millar AB. Vascular endothelial growth factor (VEGF) in inflammatory and malignant pleural effusions. Thorax. 1999 Aug;54(8):707-10. doi: 10.1136/thx.54.8.707. PMID 10413724
- [Background] Wessel MM, Nair N, Aaker GD, Ehrlich JR, D'Amico DJ, Kiss S. Peripheral retinal ischaemia, as evaluated by ultra-widefield fluorescein angiography, is associated with diabetic macular oedema. Br J Ophthalmol. 2012 May;96(5):694-8. doi: 10.1136/bjophthalmol-2011-300774. Epub 2012 Mar 15. PMID 22423055
- [Derived] Babiuch AS, Conti TF, Conti FF, Silva FQ, Rachitskaya A, Yuan A, Singh RP. Diabetic macular edema treated with intravitreal aflibercept injection after treatment with other anti-VEGF agents (SWAP-TWO study): 6-month interim analysis. Int J Retina Vitreous. 2019 Jul 23;5:17. doi: 10.1186/s40942-019-0167-x. eCollection 2019. PMID 31367468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Early Treatment Diabetic Retinopathy Study (ETDRS) letters scores [Mean (Full Range); unit: letters]
  Study Eye | 69.95 [60 to 81]
  Fellow Eye | 73.65 [37 to 85]
Optical Coherence Tomography (OCT) - Central Subfield Thickness (CST) [Mean (Full Range); unit: µm] | 419 [328 to 585]
OCT - Cube Volume [Mean (Full Range); unit: mm3] | 11.5 [9.1 to 13.9]
OCT - Average Thickness [Mean (Full Range); unit: µm] | 300.2 [246 to 345]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Treatment Outcomes by Change in Visual Acuity From Baseline
Description: Subjects were evaluated for efficacy by the change in best corrected visual acuity from baseline.
  Best Corrected Visual Acuity (BCVA) was measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters. More letters read correctly results in a higher letter score, which represents better visual acuity.
Time Frame: Baseline and 12 months
Measure: Mean (Full Range); unit: letters
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 20
letters
  Baseline | 69.95 [60 to 81]
  12 Months | 74 [56 to 85]

2. Primary Outcome: Mean Absolute Change on Central Foveal Thickness
Description: Mean absolute Central Foveal Thickness change from baseline at month 12 as measured by Spectral Domain Optical Coherence Tomography (SD-OCT), defined as the average thickness within the central 1 mm subfield of the central retina.
  Thicker measures can represent more macular edema
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: μm
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 20
μm
  Baseline | 419.7 (92)
  12 months | 287.2 (80.2)

3. Secondary Outcome: Mean Change on Visual Acuity Score
Description: The mean change from baseline in best-corrected visual acuity score at months 6,12 and 24.
  Best Corrected Visual Acuity was measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters. More letters read correctly results in a higher letter score, which represents better visual acuity.
Time Frame: Baseline, 6 months, 12 months, 24 months
Population: A total of 20 participants were enrolled; 20 completed 6 and 12 months and 16 completed the study (24 months)
Measure: Mean (Full Range); unit: letters
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 20
letters
  Baseline | 69.95 [66 to 74]
  6 months | 71.5 [54 to 83]
  12 months | 74 [56 to 85]
  24 months: number analyzed (Participants) | 16
  24 months: number analyzed (Eyes) | 16
  24 months | 75 [71 to 80]

4. Other Pre Specified Outcome: Optical Coherence Tomography (OCT) Perfusion
Description: Change in macular OCT perfusion (whole deep capillary perfusion density) at months 12 and 24 by OCT angiography
Time Frame: Baseline, 12 months,and 24 months
Population: A total of 20 participants were enrolled; 20 completed the 12 months and 16 completed the study (24 months). 15 OCT angiography out of 16 that completed the study were available for the 24-month analysis.
Measure: Mean (95% Confidence Interval); unit: percentage perfusion density
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 20
percentage perfusion density
  Baseline | 50.82 [48.63 to 53.01]
  12 months | 47.6 [45.38 to 49.87]
  24 months: number analyzed (Participants) | 15
  24 months: number analyzed (Eyes) | 15
  24 months | 46.40 [43.88 to 48.92]

5. Other Pre Specified Outcome: Number of Participants With Diabetic Retinopathy (DR) Classified by Severity
Description: The diabetic retinopathy severity changes from baseline at months 6 and 12. DR severity was judged clinically at the fundus examination.
Time Frame: Baseline, 6 months, and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Participants
  Baseline: Mild nonproliferative diabetic retinopathy (NPDR) | 0
  Baseline: Moderate NPDR | 9
  Baseline: Severe NPDR | 5
  Baseline: Proliferative diabetic retinopathy (PDR) | 6
  6 Months: Mild nonproliferative diabetic retinopathy (NPDR) | 0
  6 Months: Moderate NPDR | 9
  6 Months: Severe NPDR | 5
  6 Months: Proliferative diabetic retinopathy (PDR) | 6
  12 Months: Mild nonproliferative diabetic retinopathy (NPDR) | 2
  12 Months: Moderate NPDR | 7
  12 Months: Severe NPDR | 5
  12 Months: Proliferative diabetic retinopathy (PDR) | 6

6. Other Pre Specified Outcome: Retinal Vascular Changes by OCT Angiography
Description: Capillary Perfusion Density change at month 12 and month 24 by OCT angiography.
Time Frame: Baseline, 12 months, and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage perfusion density
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 20
percentage perfusion density
  Baseline : Super - Whole | 45.98 [43.76 to 48.21]
  Baseline : Super - Fovea | 31.15 [28.03 to 34.26]
  Baseline : Super - Parafovea | 47.34 [44.89 to 49]
  Baseline : Deep - Whole | 50.82 [48.63 to 53.01]
  Baseline : Deep - Fovea | 24.56 [20.34 to 28.77]
  Baseline : Deep - Parafovea | 53.71 [51.30 to 56.11]
  12 Months : Super - Whole | 43.56 [41.29 to 45.83]
  12 Months : Super - Fovea | 24.30 [21.11 to 27.49]
  12 Months : Super - Parafovea | 45.08 [42.58 to 47.58]
  12 Months : Deep - Whole | 47.63 [45.38 to 49.87]
  12 Months : Deep - Fovea | 24.92 [20.61 to 29.24]
  12 Months : Deep - Parafovea | 49.88 [47.42 to 52.35]
  24 Months : Super - Whole: number analyzed (Participants) | 15
  24 Months : Super - Whole: number analyzed (Eyes) | 15
  24 Months : Super - Whole | 40.68 [38.17 to 43.19]
  24 Months : Super - Fovea: number analyzed (Participants) | 15
  24 Months : Super - Fovea: number analyzed (Eyes) | 15
  24 Months : Super - Fovea | 18.51 [14.94 to 22.08]
  24 Months : Super - Parafovea: number analyzed (Participants) | 15
  24 Months : Super - Parafovea: number analyzed (Eyes) | 15
  24 Months : Super - Parafovea | 42.93 [40.24 to 45.61]
  24 Months : Deep - Whole: number analyzed (Participants) | 15
  24 Months : Deep - Whole: number analyzed (Eyes) | 15
  24 Months : Deep - Whole | 46.40 [43.88 to 48.92]
  24 Months : Deep - Fovea: number analyzed (Participants) | 15
  24 Months : Deep - Fovea: number analyzed (Eyes) | 15
  24 Months : Deep - Fovea | 23.69 [18.87 to 28.50]
  24 Months : Deep - Parafovea: number analyzed (Participants) | 15
  24 Months : Deep - Parafovea: number analyzed (Eyes) | 15
  24 Months : Deep - Parafovea | 48.83 [46.08 to 51.58]

7. Other Pre Specified Outcome: Foveal Avascular Zone (FAZ) Changes
Description: FAZ Area change at month 12 and month 24 by OCT angiography.
Time Frame: Baseline, 12 months, and 24 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: mm2
Units Other Than Participants: Eyes
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 20
mm2
  Baseline | 0.30 [0.22 to 0.37]
  12 Months | 0.34 [0.27 to 0.41]
  24 Months: number analyzed (Participants) | 15
  24 Months: number analyzed (Eyes) | 15
  24 Months | 0.40 [0.33 to 0.48]

8. Other Pre Specified Outcome: Number of Participants With Absence of Retinal Fluid as Measured by OCT
Description: The percentage of participants that were considered anatomically 'dry' by SDOCT at months 6 and 12 and transitioned to the every-8-weeks treatment regimen.
Time Frame: Baseline, 6 months, and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 20
Participants
  Baseline: every-4-weeks regimen | 20
  Baseline: every-8-weeks regimen | 0
  6 Months: every-4-weeks regimen | 13
  6 Months: every-8-weeks regimen | 7
  12 Months: every-4-weeks regimen | 5
  12 Months: every-8-weeks regimen | 15

9. Other Pre Specified Outcome: Number of Participants That Gained or Lost Letters of Visual Acuity.
Description: The percentage of participants who gained or lost 5, 10, and 15 letters or more of vision at month 12.
  Visual Acuity (BCVA) was measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score starting at 4 meters.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 20
percentage of participants
  Lost 15 letters | 5
  Lost 14 to 10 letters | 5
  Lost 9 to 5 letters | 10
  Lost 1 to 4 letters | 5
  Gained 0 to 4 letters | 30
  Gained 5 to 9 letters | 10
  Gained 10 to 14 letters | 25
  Gained more than 15 letters | 10

ADVERSE EVENTS:
Time Frame: 24 months
Description: Safety evaluations included ocular and non-ocular events reported by patients during or between study visits. Adverse Events (AE) could also be detected through assessment and were recorded in case report forms. AEs were categorized according to severity (mild, moderate or severe) and relationship to study drug (related/not related).
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=20)
Hypertension and Hyperglycemia (General disorders) | 1 (1) — Patient with hypertension hyperglycemia requiring hospitalization. Categorized as unrelated to the study drug.
Chest pain (Cardiac disorders) | 1 — Chest pain requiring cardiac catheterization. Categorized as unrelated to the study drug.
Bilateral lower limb cellulitis (Infections and infestations) | 1 — Cellulitis requiring hospitalization. Categorized as unrelated to the study drug.
Death of unknown cause (General disorders) | 1 — Patient died to unrelated causes from study

LIMITATIONS AND CAVEATS:
Limitations of this study include its small sample size, lack of non-transitioned comparison group, and lack of standardization of other anti-vascular endothelial growth factors (anti-VEGF) therapies prior to trial initiation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT02559180/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT02559180/SAP_001.pdf